CLINICAL TRIAL: NCT00090116
Title: A Randomized, Double-Blind,Placebo-Controlled Evaluation of the Safety and Efficacy of Neramexane Monotherapy in Patients With Moderate to Severe Dementia of the Alzheimer's Type
Brief Title: The Safety and Efficacy of Neramexane in Patients With Moderate to Severe Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NER-MD-02
Record Dates: First submitted 2004-08-24; First posted 2004-08-26 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Alzheimer's Disease
Keywords: Neramexane; NMDA receptor antagonist; Memory Loss; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease; Memory Disorders | interventions — neramexane

INTERVENTIONS:
Drug: Neramexane

SUMMARY:
Memory loss and difficulties with thinking associated with Alzheimer's disease may be due to chronic release of a brain chemical called glutamate. Glutamate helps transmit messages between nerve cells through interaction with a certain type of receptor (N-methyl-D-aspartate, NMDA) on the cell. Neramexane is a new drug that blocks the effects of excessive glutamate at the receptor (NMDA receptor antagonist).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe Alzheimer's disease;
* ambulatory patients

Exclusion Criteria:

* folate deficiency;
* clinically significant central nervous system disease other than Alzheimer's disease;
* clinically significant pulmonary, gastrointestinal, renal, hepatic, endocrine or cardiovascular disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2003-03; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Pivotal Research Centers, Peoria, Arizona
  - 21st Century Neurology, Phoenix, Arizona
  - Margolin Brain Institute, Fresno, California
  - Pharmacology Research Institute, Northridge, California
  - UCI Medical Center, Orange, California
  - Pacific Research Network, San Diego, California
  - Affiliated Research Institute, San Diego, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Baumel-Eisner Neuromedical Institute, Fort Lauderdale, Florida
  - Berma Research Group, Hialeah, Florida
  - Palm Beach Neurological Center, Palm Beach Gardens, Florida
  - Neurology Clinical Research, Inc., Plantation, Florida
  - University of South Florida, Tampa, Florida
  - Palm Beach Neurology, West Palm Beach, Florida
  - Indiana Universisty Medical Center, Indianapolis, Indiana
  - Lexington Clinic, Lexington, Kentucky
  - J. Gary Booker, MD, Shreveport, Louisiana
  - Mood and Memory Clinic of Michigan, Farmington Hills, Michigan
  - St. Louis University, St Louis, Missouri
  - Alzheimer's Research Corporation, Lakehurst, New Jersey
  - Joel Ross, MD, Long Branch, New Jersey
  - Ubhc/Umdnj, Piscataway, New Jersey
  - Upstate Clinical Research, Albany, New York
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York
  - Monroe Community Hospital, Rochester, New York
  - Behavioral Medical Research of Saten Island, PC, Staten Island, New York
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Neurology and Neuroscience Center of Ohio, Toledo, Ohio
  - Summit Research Network, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - North Texas Neurology Research, Wichita, Texas
  - Pioneer Pharmaceutical Research, Midvale, Utah

REFERENCES:
- See also: Related Info — http://www.alzheimers.org